CLINICAL TRIAL: NCT06512454
Title: Prospective Observational Study on the Natural History of Alpha-1 Antitrypsin Deficiency and Associated Liver Disease
Brief Title: A Study in Adults to Learn About Inherited Alpha-1 Antitrypsin Deficiency (AATD) and AATD Related Liver Problems
Acronym: ALPHATUDE
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-999-5008
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Alpha1-Antitrypsin Deficiency
Keywords: Drug Therapy
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: AATD-Pi*ZZ Genotype/Phenotype: Participants who have been diagnosed with Alpha-1 Antitrypsin Deficiency homozygote ZZ (AATD-Pi*ZZ) genotype/phenotype with mild or without liver disease manifestations will be enrolled and data will be prospectively collected per routine care throughout the follow-up period.
  Interventions: Other: No Intervention
- Cohort 2: AATD-Pi*SZ Genotype/Phenotype: Participants who have been diagnosed with alpha-1 antitrypsin deficiency heterozygous SZ (AATD-Pi*SZ) genotype/phenotype with moderate-advanced or severe liver disease manifestations will be enrolled and data will be prospectively collected per routine care throughout the follow-up period.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The main aim of this study is to learn about liver problems caused by the lack of alpha-1 antitrypsin (called Alpha-1 Antitrypsin Deficiency or AATD) in adults when not treated (this is called the natural history of a condition) over 5 years. Other aims are to learn what can predict the AATD-liver condition starting and getting better or worse, describe how this condition is currently being diagnosed and watched in normal hospital care, and describe how the AATD also affects and adult's lung function.

Data in this study will be collected to include medical history of a participant, including the date AATD was first identified and/or the date on which the first AATD-related liver or lung problems were diagnosed. At study start and then every year until study end, participants will be asked to completed questionnaires (called patient-reported outcomes or PRO).

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all the following criteria will be included in the study.

Cohorts 1 and 2:

1. Willing to provide written informed consent or currently enrolled in an ongoing participating AATD patient registry that does not require reconsenting to participate in the study.
2. >=18 years of age at enrollment in this study.
3. Participants with documented diagnosis of AATD, meeting the following criteria:

   1. Cohort 1 (AATD-Pi*ZZ genotype/phenotype).

      • Pi*ZZ genotype as documented from rapid genetic assay, sequencing, or polymerase chain reaction (PCR), or Pi*ZZ phenotype as documented from iso-electric focusing (IEF) electrophoresis.
   2. Cohort 2 (AATD-Pi*SZ genotype/phenotype with liver disease manifestation).

      * Pi*SZ genotype as documented from rapid genetic assay, sequencing, or PCR, or Pi*SZ phenotype as documented from IEF electrophoresis, and
      * Moderate-advanced or severe liver disease manifestation as defined by either liver biopsy or surrogate laboratory or imaging measures, as determined through:

        * Lab and imaging measures to define liver disease manifestation

Exclusion Criteria:

Participants who meet any following criteria will be excluded from the study.

1. Documented AATD genotype/phenotype other than Pi*ZZ or Pi*SZ.
2. History of liver transplant.
3. No results for either biopsies, magnetic resonance elastography (MRE), fibro scan (vibration controlled transient elastography [VCTE]), or Aspartate aminotransferase to platelet ratio index (APRI) in the 24 months prior to the index/enrollment date and has none of these tests ordered during the index period.
4. Participants who had previously been treated or in an active participation in an interventional trial studying liver or lung disease.
5. Treatment with liver directed AATD investigational therapy as part of a compassionate use request.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have already been diagnosed with AATD of genotype/phenotype Pi*ZZ, with mild or without liver disease manifestation, or with genotype/phenotype of Pi*SZ with moderate-advanced or severe liver disease manifestation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2032-04-06 (Estimated); Study Completion 2032-04-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Liver Disease Progression | Baseline up to 5 years
  Liver disease progression will be defined as advancement in greater than or equal to (>=1) fibrosis stage: example any progression from fibrosis stage (F)0 to F1, F1 to F2, F2 to F3 etc. and/or occurrence of any of these composite events: a) advancement in >=1 fibrosis stage, b) development of a liver disease-related clinical event, c) model for end-stage liver disease (MELD) score increase, or d) receipt of a liver transplant MELD score increase, or d) receipt of a liver transplant. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis. The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome.
Time to Liver Disease Progression | Baseline up to 5 years
  Time to liver disease progression is defined as time to advancement in >=1 fibrosis stage (example F1 to F2, F2 to F3 etc.) and/or time to the earliest of: Advancement in >=1 fibrosis stage, or development of a liver disease-related clinical event, or MELD score increase or receipt of a liver transplant. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis. The MELD score ranges from 6 to 40 with higher scores indicating more severe liver disease and a worse outcome.
Time to Liver Disease Trajectory | Baseline up to 5 years
  Time to liver disease trajectory is defined as time of transition from F0/F1 to F2, F2 to F3, F3 to F4, F4 to the decompensating event or liver transplant and first to second decompensating event and all subsequent decompensating events or liver transplant. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis.
Probability of Transition in Liver Disease Trajectory | Baseline up to 5 years
  Probability of liver disease trajectory is defined as probability of transition from F0/F1 to F2, F2 to F3, F3 to F4, F4 to the decompensating event or liver transplant and first to second decompensating event and all subsequent decompensating events or liver transplant. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis.
Percentage of Participants With Disease Regression | Baseline up to 5 years
  Disease regression is defined as decrease in >=1 fibrosis staging. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis.
Time to Liver Disease Regression | Baseline up to 5 years
  Time to liver disease regression is defined as time to decrease in >=1 fibrosis stage. The fibrosis stages range from F0 to F4, with F0 indicating no fibrosis and F4 indicating cirrhosis.
Percentage of Participants With All-cause Mortality and Cause-specific Mortality | Baseline up to 5 years
  Cause-specific mortality is defined as mortality due to liver failure or complications of cirrhosis/portal hypertension or hepatocellular carcinoma, or infections secondary to liver failure.
Time to Death (All-causes) and Cause-specific Death (Liver Disease-specific Causes) | Baseline up to 5 years
  Cause-specific mortality is defined as mortality due to liver failure or complications of cirrhosis/portal hypertension or hepatocellular carcinoma, or infections secondary to liver failure.

SECONDARY OUTCOMES:
Percentage of Participants Who Develop Lung Disease | Baseline up to 5 years
  Development of lung disease will be defined as either a forced expiratory volume in 1 second (FEV1) percent (%) predicted of less than (<) 70% or the diagnosis of at least 1 lung condition (chronic obstructive pulmonary disease [COPD], emphysema, bronchiectasis, chronic bronchitis).
Proportion of Participants With Lung Disease at Baseline who Experience Lung Disease Progression at 5 Years | Baseline up to 5 years
  Lung disease progression is defined as changes in pulmonary function (defined as >=10% absolute change in FEV1, forced vital capacity [FVC], or diffusing capacity of the lungs for carbon monoxide [DLCO]).
Number of Participants With Invasive and Non-Invasive Assessment for Liver Disease | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- University of Florida, Gainesville, Florida, United States
- Universitätsklinikum Aachen AöR, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/8eac08f5b4464a1d??page=1&idFilter=TAK-999-5008